CLINICAL TRIAL: NCT06176287
Title: Assessment of Pain Associated With Insertion Torque and Correlation of Primary Implant Stability Measurement Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Collaborators: MIS Implant Technologies, Ltd (Industry)
Responsible Party: Principal Investigator, Mehmet Gumus Kanmaz, DDS, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-3.2/9
Record Dates: First submitted 2023-10-09; First posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Dental Implantation
Keywords: dental implants; dental implantation; pain assessment
MeSH Terms: interventions — Dental Implantation

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High insertion torque group (Active Comparator): Fifteen patients (eight females and seven males) with a single-tooth deficiency bilaterally in the molar region of the lower jaw were included in the study. Implant placement with high insertion torque was planned on one side of the jaw. The implant drills were applied as recommended by the company. To achieve high insertion torque, the single-use final drill from the implant box was not used in the high torque group.
  Interventions: Procedure: Dental Implantation with high torque
- Low insertion torque group (Active Comparator): Fifteen patients (eight females and seven males) with a single-tooth deficiency bilaterally in the molar region of the lower jaw were included in the study. Implant placement with low insertion torque was planned on the otherside of the jaw. The implant drills were applied as recommended by the company. To achieve low insertion torque, the single-use final drill was applied two times.
  Interventions: Procedure: Dental Implantation with low torque

INTERVENTIONS:
Procedure: Dental Implantation with high torque — Fifteen patients with bilateral single-tooth loss in the posterior mandible will be included in the study. One implant was randomly placed with high insertion torque in each patient. A total of 15 implants will be placed, and insertion torque values will be recorded.
  Arms: High insertion torque group
Procedure: Dental Implantation with low torque — Fifteen patients with bilateral single-tooth loss in the posterior mandible will be included in the study. One implant was randomly placed with low insertion torque in each patient. A total of 15 implants will be placed, and insertion torque values will be recorded.
  Arms: Low insertion torque group

SUMMARY:
The objective of this observational study is to evaluate the primary stability of dental implants and the relationship between insertion torque and patients' pain levels assessed with the visual analogue scale (VAS)

DETAILED DESCRIPTION:
Primary implant stability plays a key role in providing osseointegration. Higher insertion torque indicates higher primary stability. However, the effect of increased insertion torque on patient pain levels has not been clearly demonstrated. Several methods for measuring primary stability have been defined so far. Insertion torque, periotest measurements, and resonance frequency analysis are mostly preferred due to their ease of use and non-invasiveness.

The aim of the present study is to evaluate the relationship between insertion torque and patients' pain levels assessed with the visual analogue scale (VAS) and to assess the relationship between insertion torque, periotest measurements, and resonance frequency analysis.

ELIGIBILITY:
Inclusion Criteria:

* No contraindications for implant surgery;
* Bilateral single-tooth loss in the posterior mandible;
* Sufficient bone amount for implant diameter and height at the implant site;
* At least 3 months after tooth extraction at the implant site;

Exclusion Criteria

* History of chronic infection or pain at the implant site;
* History of radiotherapy to the head and neck region for any reason;
* Local or systemic causes of persistent anti-inflammatory or analgesic medication;
* Patients with suspicion of pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-04-19 (Actual); Primary Completion 2016-09-09 (Actual); Study Completion 2016-10-14 (Actual)

PRIMARY OUTCOMES:
Pain levels assessed with the visual analogue scale (VAS) | 7 days
  Patients will be asked to record the number of painkillers taken each day and evaluate their pain levels using a 0-10 VAS form before and after the operation. A score of 0 indicated no pain while 10 indicated the worst pain possible. A VAS score of 1-3 indicated mild pain, 4-6 indicated moderate pain, and 7-10 indicated very severe pain.

SECONDARY OUTCOMES:
Insertion torque values | 1 day
  After the implant slots were prepared, the coronal part of the implants (MIS Implant Technologies, Bar Lev Industrial Park, Israel) were placed into the slots at 25 rpm without irrigation until the coronal part was at the same level with the ridge top. The maximum insertion torque was recorded while the implants were placed with the help of a physiodispenser that can measure the insertion torque (Kavo Expertsurg lux physiodispenser, KaVo Dental GmbH, Biberach, Germany).
Periotest measurements | 1 day
  Measurements were made with the Periotest (Siemens AG, Bensheim, Germany) device and recorded as PTV (perio test value).
Resonance frequency analysis values | 1 day
  A SmartPeg (Integration Diagnostics AB; Gothenburg, Sweden) suitable for the implant was attached to measure primary implant stability with radiofrequency. Radiofrequency analysis was performed in both mesiodistal and buccolingual directions with the Osstell Mentor (Integration Diagnostics AB; Gothenburg, Sweden) device and the measurements were recorded.